CLINICAL TRIAL: NCT06022328
Title: Impact of Epigenetic Age on Clinic-biological Presentation and Prognosis in Myeloproliferative Neoplasms Epigenetic Age in Myeloproliferative Neoplasms (EpiC)
Acronym: EpiC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/15
Record Dates: First submitted 2023-07-24; First posted 2023-09-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Myeloproliferative Neoplasm
Keywords: Myeloproliferative Neoplasm; Epigenetic age; Thrombosis; Myelofibrosis; Leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombosis; Primary Myelofibrosis; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with ET: 45 patients with ET:
  * 15 without thrombotic event (neither at diagnosis nor during follow-up)
  * 15 with thrombotic events (thrombosis at diagnosis or within 2 years of diagnosis)
  * 15 who progressed to myelofibrosis or AML during follow-up
  Interventions: Biological: Assessment of the epigenetic age
- Patients with PV: 45 patients with PV
  * 15 without thrombotic event (neither at diagnosis nor during follow-up)
  * 15 with thrombotic event (thrombosis at diagnosis or within 2 years of diagnosis)
  * 15 who progressed to myelofibrosis or AML during follow-up
  Interventions: Biological: Assessment of the epigenetic age
- Patients with PMF: 20 patients with PMF:
  * 10 without transformation into AML
  * 10 patients who progressed to AML
  Interventions: Biological: Assessment of the epigenetic age
- Patients without MPN: 10 patients without MPN
  Interventions: Biological: Assessment of the epigenetic age

INTERVENTIONS:
Biological: Assessment of the epigenetic age — Retrospective assessment of the epigenetic age on DNA samples obtained at diagnosis

SUMMARY:
Myeloproliferative Neoplasms (MPN) are hematological malignancies characterized by the excessive production of myeloid cells. MPN can be complicated by thrombosis and evolution into more aggressive diseases (myelofibrosis and acute leukemia). Aging remains the principal factor determining patients' survival in MPN. In recent years, DNA methylation has appeared as a mean to measure aging via the development of epigenetic clocks that have also been associated with the occurrence of thrombosis and cancer. The epiC project aims at determining epigenetic age of MPN patients and search for an association between this parameter and thrombotic/hematological complications.

DETAILED DESCRIPTION:
Myeloproliferative Neoplasia (MPN) are hematological malignancies characterized by the excessive production of myeloid cells. They include Essential Thrombocythemia (ET), Polycythemia Vera (VP) and Primary Myelofibrosis (PMF). Thrombosis are the most frequent complications and are largely responsible for the morbidity and mortality observed in ET and PV patients. The most feared complications are hematological transformations (into myelofibrosis for PV and ET, into acute myeloid leukemia for PV, ET and PMF). The prognostic assessment of MPN patients is mainly based on clinical data. Although recent studies have shown that certain mutations are associated with a poorer prognosis, age remains the main risk factor affecting survival in MPN patients. Recent studies have shown that DNA methylation can be used to determine an "epigenetic age". Interestingly, this epigenetic age is associated with the development of cardiovascular disease and cancer.

In this project, the epigenetic age of MPN patients will be determined by studying the DNA methylation at diagnosis using the Infinium Human MethylationEPIC kit (Illumina). Epigenetic age will be determined with the most commonly used epigenetic clocks (DNAmAge, DNAmHannum, DNAmPhenoAge, DNAmSkinClock, DNAmGrimAge, intrinsic epigenetic age acceleration, extrinsic epigenetic age acceleration). It will be searched for an association between accelerated epigenetic aging (as assessed by the difference between epigenetic age and chronological age) and the type of MPN, the clinical and biological presentation at diagnosis (including the mutational profile of patients) and the occurrence of thrombosis and hematological evolution into myelofibrosis and/or acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

For the 110 patients with MPN:

* Patients with PV, ET or PMF
* DNA extracted from purified granulocytes at time of diagnosis
* No treatment likely to impact DNA methylation (chemotherapy, immunosuppressants in particular)

For the 10 subjects without MPN:

* Absence of hematological malignancy
* Search for JAK2V617F mutation in the context of reactive thrombocytosis or secondary polycythemia
* Absence of treatment likely to impact DNA methylation (chemotherapy, immunosuppressants in particular)

Exclusion Criteria:

For the 110 patients with MPN:

* Patients without PV, ET or PMF
* Patients without purified granulocytes DNA available at time of diagnosis
* Patients treated by cytoreductive drug, demethylating agent, chemotherapy or immunosuppressive therapy at the time of DNA sampling
* Patients with less than 2 years' follow-up

For the 10 subjects in NMP :

* Patients with hematological malignancy and/or solid cancer
* Patients treated by cytoreductive drug, demethylating agent, chemotherapy or immunosuppressive therapy at the time of DNA sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Myeloproliferative Neoplasia (MPN) : Essential Thrombocythemia (ET), Polycythemia Vera (VP) or Primary Myelofibrosis (PMF)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Accelerated ageing of patients | At inclusion, up to 1 year after diagnosis
  Accelerated ageing will be defined as an increased difference between the epigenetic age (calculated from DNA methylation data with the different molecular clocks described: DNAmAge, DNAmHannum, DNAmPhenoAge, DNAmSkinClock, DNAmGrimAge, intrinsic epigenetic age acceleration, extrinsic epigenetic age acceleration) and the chronological age

SECONDARY OUTCOMES:
Type of MPN (ET, PV or PMF) at diagnosis | At inclusion, up to 1 year after diagnosis
  We will study patients with a diagnosis of ET, PV or PMF as defined by the WHO classification of hematological malignancies
Transformation into secondary myelofibrosis or acute leukemia | From date of inclusion until documentation of the event, assessed up to 5 years
  Evolution toward secondary myelofibrosis or acute leukemia will be defined according to the WHO classification of hematological malignancies
Occurrence of thrombosis prior to diagnosis or during follow-up of the disease | Between 1 year before and 2 years after MPN diagnosis
  Occurrence of myocardial infarction, ischemic stroke, deep vein thrombosis, pulmonary embolism, splanchnic thrombosis or any other significant thrombosis. Tinnitus, vertigo, headaches, erythromelalgia as well as superficial vein thrombosis will not be considered as thrombotic events
Leukocytes | At inclusion, up to 1 year after diagnosis
  Leukocytes level on blood count in G/L
Platelets | At inclusion, up to 1 year after diagnosis
  Platelet level on blood count in G/L
Granulocytes | At inclusion, up to 1 year after diagnosis
  Granulocytes level on blood count in G/L
Monocytes | At inclusion, up to 1 year after diagnosis
  Monocytes level on blood count in G/L
Hemoglobin | At inclusion, up to 1 year after diagnosis
  Hemoglobin level on blood count in g/dL
Hematocrit | At inclusion, up to 1 year after diagnosis
  Hematocrit level on blood count in %
Additional somatic mutation | At inclusion, up to 1 year after diagnosis
  In up to 50% of MPN patients, genetic variants can be detected in genes such as DNMT3A, TET2, ASXL1, SRSF2, SF3B1, U2AF1, EZH2 or TP53. We will determine which somatic genetic variant is detected by high throughput sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, service Hématologie Biologique, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No